CLINICAL TRIAL: NCT07376889
Title: COMBAT-SAB: Combination Antibiotic Therapy for Staphylococcus Aureus Bacteremia
Brief Title: Combination Antibiotic Therapy for Staphylococcus Aureus Bacteremia
Acronym: COMBAT-SAB
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Brandon Webb, Associate Professor of Research, Division of Infectious Diseases, Intermountain Health Care, Inc.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1053331
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Staphylococcus Aureus Bacteremia
Keywords: Combination antibiotic therapy

STUDY DESIGN:
Intervention Model Description: Platform, embedded, pragmatic clinical trial using a multiple-crossover cluster-randomized design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with methicillin-sensitive S. aureus bacteremia (MSSAB) (Experimental): Patients with methicillin-sensitive S. aureus bacteremia (MSSAB) will be assigned to one of two different antibiotic treatment strategies appropriate for MSSA: 1) antibiotic monotherapy, or 2) combination antibiotic therapy
  Interventions: Drug: Antibiotic Monotherapy (AM) for patients with methicillin-sensitive S. aureus bacteremia (MSSAB); Drug: Combination Antibiotic Therapy (CAT) for patients with methicillin-sensitive S. aureus bacteremia (MSSAB)
- Patients with methicillin-resistant S. aureus bacteremia (MRSAB) (Experimental): Patients with methicillin-resistant S. aureus bacteremia (MRSAB) will be assigned to one of two different antibiotic treatment strategies appropriate for MRSA: 1) antibiotic monotherapy, or 2) combination antibiotic therapy
  Interventions: Drug: Antibiotic Monotherapy (AM) for patients with methicillin-resistant S. aureus bacteremia (MRSAB); Drug: Combination Antibiotic Therapy (CAT) for patients with methicillin-resistant S. aureus bacteremia (MRSAB)

INTERVENTIONS:
Drug: Antibiotic Monotherapy (AM) for patients with methicillin-sensitive S. aureus bacteremia (MSSAB) — Intravenous anti-staphylococcal beta-lactam, either cefazolin or nafcillin, per the discretion of the treating physician.
  Arms: Patients with methicillin-sensitive S. aureus bacteremia (MSSAB)
Drug: Antibiotic Monotherapy (AM) for patients with methicillin-resistant S. aureus bacteremia (MRSAB) — Vancomycin or daptomycin, per discretion of the treating physician
  Arms: Patients with methicillin-resistant S. aureus bacteremia (MRSAB)
Drug: Combination Antibiotic Therapy (CAT) for patients with methicillin-sensitive S. aureus bacteremia (MSSAB) — Patients with methicillin-sensitive S. aureus bacteremia (MSSAB) and no contraindications will receive an anti-staphylococcal beta-lactam, either cefazolin or nafcillin, plus ertapenem
  Arms: Patients with methicillin-sensitive S. aureus bacteremia (MSSAB)
Drug: Combination Antibiotic Therapy (CAT) for patients with methicillin-resistant S. aureus bacteremia (MRSAB) — Daptomycin plus ceftaroline
  Arms: Patients with methicillin-resistant S. aureus bacteremia (MRSAB)

SUMMARY:
The purpose of this study is to see if, in selected patients with a serious bacterial infection of the bloodstream, treating the bacterial infection with a combination of antibiotics is more effective than treating the infection with a single antibiotic. Participants must have blood cultures which are positive for a certain type of bacteria.

DETAILED DESCRIPTION:
Staphyloccocus aureus bacteremia (SAB) is a common infectious disease condition in hospitalized patients which is associated with significant morbidity, excessive costs, and high mortality, despite effective antibiotic therapy. This pragmatic study is designed to test the hypothesis that outcomes in adults hospitalized with SAB will be improved by using combination antibiotic therapy (CAT) as early, targeted therapy in a high-risk subgroup. A group of patients identified early in their course as meeting at least one high-risk criterion who have no contraindications will be treated with one of two antibiotic strategies commonly used within usual care, namely: 1) antibiotic monotherapy or 2) combination antibiotic therapy, depending on the random assignment for each hospital, each month. Low-risk patients will be treated per usual care. Data from all patients admitted to participating hospitals with SAB will be included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Alive and admitted to an Intermountain Health (IH) hospital acute care unit at enrollment
* Initial positive blood culture with either methicillin-resistant Staphylococcus aureus (MRSA) or methicillin-susceptible Staphylococcus aureus (MSSA), collected:

  1. on or during the index admission to an IH hospital, or
  2. in an ambulatory setting (laboratory, clinic or emergency department) within 48 hours of the index admission, or
  3. at a non-IH network hospital within 24 hours of subsequent transfer to an IH hospital

     Exclusion Criteria:
* Patient requests that patient health data not be included in the analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2096 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Desirability of Outcome Ranking (DOOR) | From enrollment to 30 days post enrollment
  The DOOR ordinal scale includes four possible outcomes: treatment failure, infectious complications, antibiotic-associated adverse events and death. The ordinal scale comprises five levels: levels 1-4 are defined by survival at 30 days and the presence of either none, one, two or three of three possible outcomes; level 5 indicates death before 30 days. A DOOR analysis estimates the probability that overall outcomes in any given subject in one group are overall superior to those in a random subject from the other treatment group; probabilities >50% reject the null hypothesis.

SECONDARY OUTCOMES:
90-day hospital-free days alive | From enrollment to 90 days after enrollment
  Number of days the patient is alive and out of the hospital
30-day all cause mortality | From enrollment to 30 days after enrollment
  Number of deaths from any cause within 30 days after enrollment
90-day all-cause mortality | From enrollment to 90 days after enrollment
  Number of deaths from any cause within 90 days after enrollment
30-day bacteremia-free days | From enrollment to 30 days after enrollment
  Number of days without bacteremia within 30 days after enrollment
Length of stay | Measured at the time of hospital discharge, up to 30 days after enrollment
  Number of days in the hospital following enrollment
Total hospital direct costs | Measured at the time of hospital discharge, up to 30 days after enrollment
  Total financial charges incurred by a patient during their hospitalization
Total inpatient antibiotic cost | Measured at the time of hospital discharge, up to 30 days after enrollment
  Total cost of all antibiotics received by a patient while hospitalized
Combination antibiotic days | Measured from the time of enrollment until study day 7, death, or hospital discharge
  Number of days a patient receives combination antibiotic therapy (CAT) as defined in protocol, instead of antibiotic monotherapy (AM)
Antibiotic-associated adverse events | From enrollment to 30 days after enrollment
  Number and type of patient adverse events definitively associated with the receipt of antibiotics while hospitalized
Clostridioides difficile infection | From enrollment to 30 days after hospital discharge
  Presence of infection with Clostridioides difficile while hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Brandon J Webb, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (13):
- United States (13):
  - Platte Valley Hospital, Brighton, Colorado
  - Saint Joseph Hospital, Denver, Colorado
  - St. Mary's Regional Hospital, Grand Junction, Colorado
  - Good Samaritan Hospital, Lafayette, Colorado
  - Lutheran Medical Center, Wheat Ridge, Colorado
  - St. Vincent Regional Hospital, Billings, Montana
  - St. James Hospital, Butte, Montana
  - Holy Rosary Hospital, Miles City, Montana
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley Hospital, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - St. George Regional Hospital, St. George, Utah

IPD SHARING:
Plan to Share IPD: Yes
In order to protect patient privacy and comply with relevant regulations, identified data will be unavailable. Requests for deidentified data from qualified researchers with appropriate ethics board approvals and relevant data use agreements will be processed by the Intermountain Office of Research, officeofresearch@imail.org
Time Frame: Data sharing will be available six months after anticipated enrollment completion, estimated August 2029, for a period to be determined by the Intermountain Office of Research and IRB
Access Criteria: Will be determined on an individual basis, upon request to the IH Office of Research.